CLINICAL TRIAL: NCT02731599
Title: The Effects of Treadmill Training With Visual and Auditory Cues on Gait Parameters in Parkinsonian Patients in Advanced Stages of Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: treadmill and PD
Record Dates: First submitted 2016-04-03; First posted 2016-04-07 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; treadmill; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treadmill training (Experimental): 20-minutes treadmill training per day, 6 times a week, for 4 weeks
  Interventions: Procedure: treadmill training with cues

INTERVENTIONS:
Procedure: treadmill training with cues — 20-minutes treadmill training per day, 6 times a week, for 4 weeks. Treadmill speed was previously set at 2.0 km/h and progressively increased until a maximum of 3.5 km/h, taking always into account the patients' physical abilities. All patients were evaluated at the enrolment and at the end of the 4-weeks treatment. The first evaluation consisted in one-minute walking on treadmill without the use of cues at 1.5 km/h speed, for all patients. The outcome measurements were: the average length of the right step, the average length of the left step, the coefficient of variance of both steps, and the gait cycle.

SUMMARY:
The first aim of this study was to evaluate the effect of a gait training using treadmill with visual and auditory cues in patients in stages IV Hoehn & Yahr (H&Y). The second aim was to compare the obtained data of these patients in advanced stages with those in mild to moderate stages.

DETAILED DESCRIPTION:
Gait is altered in Parkinson's disease (PD) patients. It has been shown that treadmill training with visual and auditory cues is useful in improving the gait's parameters in patients in early-moderate stages of disease. No data are available about the effectiveness of this training in those subjects in advanced stages of PD. The first aim of this study was to evaluate the effect of a gait training using treadmill with visual and auditory cues in patients in stages IV Hoehn & Yahr (H&Y). The second aim was to compare the obtained data of these patients in advanced stages with those in mild to moderate stages.

150 patients with PD in early-moderate and advanced stages of disease (50 in H&Y stage 2, group 1, 50 in H&Y stage 3, group 2 and 50 in H&Y stage 4, group 3) were enrolled. All patients underwent an intensive treatment: 20-minutes treadmill training per day, 6 times a week, for 4 weeks. Treadmill speed was previously set at 2.0 km/h and progressively increased until a maximum of 3.5 km/h, taking always into account the patients' physical abilities. All patients were evaluated at the enrolment and at the end of the 4-weeks treatment. The first evaluation consisted in one-minute walking on treadmill without the use of cues at 1.5 km/h speed, for all patients. The outcome measurements were: the average length of the right step, the average length of the left step, the coefficient of variance of both steps, and the gait cycle.

ELIGIBILITY:
Inclusion Criteria:

Parkinson Disease

Exclusion Criteria:

comorbidity with other neurological condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Length of step | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Generale di zona Moriggia Pelascini, Gravedona Ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No